CLINICAL TRIAL: NCT05887193
Title: Effects of Contemporary Cycling Saddle Designs on Penile Transcutaneus Oxygen and Carbon Dioxide Levels in Elite Road Cyclists Riding on a Stationary Trainer
Acronym: EC-SADDLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milan Martínek (Other)
Responsible Party: Sponsor-Investigator, Milan Martínek, Mgr. Ph.D., Charles University, Czech Republic
Organization: Charles University, Czech Republic (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CharlesUCR - EC-SADDLE; UK FTVS 002/2023 (Other: aculty of Physical Education and Sport, Charles University, Ethics Committee)
Record Dates: First submitted 2023-04-21; First posted 2023-06-02 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Healthy; Cyclists; Blood Gas Monitoring, Transcutaneous; Penile Numbness
Keywords: saddle; pressure; bicycling; erectile dysfunction; hypesthesia; transcutaneous blood gas monitoring; bike fit; biothesiometry
MeSH Terms: conditions — Erectile Dysfunction; Hypesthesia | interventions — Blood Gas Monitoring, Transcutaneous; Heart Rate Determination

STUDY DESIGN:
Intervention Model Description: This study employed a randomized, within-subject, crossover design with counterbalancing to evaluate the effects of three different cycling saddles on transcutaneous penile oxygen (TcPO₂) and carbon dioxide (TcPCO₂) pressures in elite male cyclists. Participants cycled for 10 minutes on each saddle on a stationary trainer, with 5 minute rest intervals between conditions. To minimize potential order effects, participants were randomly assigned to one of six saddle-order sequences.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (Active Comparator): Order of saddle testing: Joyseat saddle - Specialized Power saddle - Fizik Tundra M5 saddle
  Interventions: Device: Biothesiometry; Device: Transcutaneous blood gas monitoring; Device: Cycling on a home trainer; Device: Bike Fitting; Device: Heart rate monitoring; Device: Velomotrik smart cover BT
- Group 2 (Active Comparator): Order of saddle testing: Joyseat saddle - Fizik Tundra M5 saddle - Specialized Power saddle
  Interventions: Device: Biothesiometry; Device: Transcutaneous blood gas monitoring; Device: Cycling on a home trainer; Device: Bike Fitting; Device: Heart rate monitoring; Device: Velomotrik smart cover BT
- Group 3 (Active Comparator): Order of saddle testing: Specialized Power saddle - Fizik Tundra M5 saddle - Joyseat saddle
  Interventions: Device: Biothesiometry; Device: Transcutaneous blood gas monitoring; Device: Cycling on a home trainer; Device: Bike Fitting; Device: Heart rate monitoring; Device: Velomotrik smart cover BT
- Group 4 (Active Comparator): Order of saddle testing: Specialized Power saddle - Joyseat saddle - Fizik Tundra M5 saddle
  Interventions: Device: Biothesiometry; Device: Transcutaneous blood gas monitoring; Device: Cycling on a home trainer; Device: Bike Fitting; Device: Heart rate monitoring; Device: Velomotrik smart cover BT
- Group 5 (Active Comparator): Order of saddle testing: Fizik Tundra M5 saddle - Joyseat saddle - Specialized Power saddle
  Interventions: Device: Biothesiometry; Device: Transcutaneous blood gas monitoring; Device: Cycling on a home trainer; Device: Bike Fitting; Device: Heart rate monitoring; Device: Velomotrik smart cover BT
- Group 6 (Active Comparator): Order of saddle testing: Fizik Tundra M5 saddle - Specialized Power saddle - Joyseat saddle
  Interventions: Device: Biothesiometry; Device: Transcutaneous blood gas monitoring; Device: Cycling on a home trainer; Device: Bike Fitting; Device: Heart rate monitoring; Device: Velomotrik smart cover BT

INTERVENTIONS:
Device: Biothesiometry — Biothesiometry using Biothesiometer (Bio Medical Instrument Co, Ohio, United States of America), placed on glans penis and second finger of nondominant hand.
  Other Names: Neurothesiometer
Device: Transcutaneous blood gas monitoring — Penile oxygen pressure using TCM5 Flex and tc84 electrode (Radiometer Medical ApS, Brønshøj, Denmark) placed on glans penis.
Device: Cycling on a home trainer — Riding a static bike Wahoo Bike (Wahoo Fitness LLC, Atlanta, Georgia, United States of America) for 3x 10 minutes in Zone 3 (Andy Coggan methodology) calculated from each individual subjects self reported Functional Threshold Power.
Device: Bike Fitting — Setting standardized posture of the rider on the bike using Retül technology (Retül, Specialized Bicycle Components Inc., Boulder, Colorado, United States of America)
Device: Heart rate monitoring — Measuring heart rate using Wahoo TICKR chest strap (Wahoo Fitness LLC, Atlanta, Georgia, United States of America)
Device: Velomotrik smart cover BT — Saddle pressure measurement, mean and max saddle pressure, saddle pressure distribution. (Velometrik GmbH, Neukieritzsch, Germany).

SUMMARY:
Aim of this research is to compare novel 3D printed cycling saddle with the bestselling saddles from two major cycling manufacturers in terms of effects on penile blood gasses and update these findings on current style of racing cycling saddles.

DETAILED DESCRIPTION:
The aim of this research is to investigate whether Posedla's 3D printed and custom-made prototype bicycle saddle Joyseat (Posedla s.r.o., Varnsdorf, Czech Republic) provide a benefit in terms of increased penile blood flow compared to the best-selling saddles from two major bicycle manufacturers. The method chosen to measure blood flow, which is commonly used in studies of this type, is referred to as transcutaneus blood gas monitoring. Measurement of TcPO2 and TcPCO2 in cyclists will be performed while riding on a cycling trainer using Radiometer TCM5 Flex (Radiometer Medical ApS, Brønshøj, Denmark) and a tc 84 electrode placed on the glans penis. Prior to the actual penile blood flow measurements, the sensitivity level of the n. pudendus (n. dorsalis penis) will be verified using biothesiometer (Bio Medical Instruments Co., Newbury, Ohio, USA), which is again commonly used in studies of this type. The pressure of the riders contact surfaces on the saddle will be evaluated with Velometrik SmartCover BT pressure mat (Velometrik GmbH, Neukieritzsch, Germany). The Wahoo KICKR Bike (Wahoo Fitness, LLC., Atlanta, Georgia, United States of America) will be used in the study, which, in addition to the possibility of individual seating adjustment, also allows to record the cyclists power and heart rate using a chest strap. The cyclists position on the bike will be measured and evaluated by infrared sensors and Retül technology (Specialized Bicycle Components, Inc., Morgan Hill, California, USA). The test will be performed using the described instrumentation in the Applied Kinesiology Laboratory at Charles University in Prague, Faculty of Physical Education and Sports and will involve riding 3x 10 minutes with 5 minutes rest in between intervals on the cycle trainer at 65-85% of the cyclists maximum individual heart rate during one visit. All measurement methods and devices are non-invasive and painless. The choice of instruments was based on their use in previously published studies of similar type and on their quality, i.e., the parameters of validity, reliability, sensitivity, specificity and availability.

ELIGIBILITY:
Inclusion Criteria:

* gender: male, age: 18-45 years, discipline: road cycling, annual mileage: more than 14000 km (Tier 3-4)

Exclusion Criteria:

* Participants other than male, diagnosed with erectile dysfunction, acute or chronic back pain, acute (especially infectious) illness or injury, and in recovery from illness or injury are not eligible for inclusion in the research

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The study design accounts only for male genitalia for the placement of the tc84 electrode.
Enrollment: 14 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2023-05-14 (Actual); Study Completion 2023-05-14 (Actual)

PRIMARY OUTCOMES:
pO2_change_point | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  Parameter pO2_change_point is the time from start of TcPO₂ measurement to the identified change point, determined within the 50-400 s interval as the transition between the fitted initial linear trend and the subsequent linear trend in TcPO₂
pCO2_change_point | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  Parameter pCO2_change_point is the time from start of TcPCO₂ measurement to the identified change point, determined within the 200-550 s interval as the transition between the fitted initial linear trend and the subsequent linear trend in TcPCO₂

SECONDARY OUTCOMES:
pO2_start | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  The value of the fitted trend at time 0 in TcPO₂ measurement.
pO2_decline | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  The slope of the fitted trend of decline in TcPO₂ after initial 20s.
pO2_end | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  The slope of the second fitted trend after pO2_change_point in TcPO₂ measurement.
pO2_part1 | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  The average value of TcPO₂ measurements in the first 20 s segment.
pO2_part2 | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  The average value of TcPO₂ measurements for the second segment, from 21 s to the trend pO2_change_point.
pO2_part3 | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  The average value of TcPO₂ measurements for the third segment after pO2_change_point.
pO2_mean | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  The average of all TcPO₂ measurements in one interval.
pO2_median | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  The median of all TcPO₂ measurements in one interval.
pCO2_start | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  The value of the fitted trend at time 0 in TcPCO₂ measurement.
pCO2_incline | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  The slope of the fitted trend of increase in TcPCO₂ in the first segment before pCO2_change_point
pCO2_end | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  The slope of the fitted trend in TcPCO₂ in the second segment after pCO2_change_point.
pCO2_part1 | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  The average value of TcPCO₂ measurements in the first segment before pCO2_change_point.
pCO2_part2 | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  The average value of TcPCO₂ measurements in the second segment after pCO2_change_point.
pCO2_mean | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  The average of all TcPCO₂ measurements in one interval.
pCO2_median | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  The median of all TcPCO₂ measurements in one interval.
logratio_11_8 | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  The logarithmic value of the ratio of the load on the front and rear parts of the saddle, where the saddle is divided in a ratio of 11:8 longitudinally.
PERI | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  Pressure value in the predefined perineal area with an area of 44 cm² in front of the ischial tuberosity maxima.
modPSRG/F | A baseline testing at the beginning of the testing protocol lasting around 5 minutes.
  Vibrotactile thresholds were measured at the volar distal phalanx of the non-dominant hand and midline of the glans penis. The probe was placed perpendicular without additional pressure. Voltage was gradually increased until the first sensation was reported, then increased further and slowly decreased until sensation was lost. Upper and lower thresholds were recorded three times per site, averaged, and used to calculate the modified Penile Sensitivity Ratio Glans/Finger via the following formula. Average of the three glans upper+lower threshold values divided by the average of the three finger upper+lower threshold values.
CVdrift | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  The percentage of cardiovascular drift calculated as a ratio between average Power and average Heart Rate between the first and second part of the 10-minute interval.
  ((P1/HR1) - (P2/HR2))/(P1/HR1) * 100 where: P1 - Average Power from first half part of the workout P2 - Average Power from second half part of the workout HR1 - Average Heart Rate from first half part of the workout HR2 - Average Heart Rate from second half part of the workout
Bike Fit parameters | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  Bike Fit values as recorded by Retül V7 System.
  KOPS - Knee Over Pedal Spindle - The fore/aft offset of the knee marker relative to the pedal spindle at 3 o'clock in the pedal stroke (90° in the downstroke) MKF - Maximum Knee Flexion - Maximum flexion of the knee joint at any point in the pedal stroke defined by the line connecting hip and knee markers and the line connecting knee and ankle markers MKE - Maximum Knee Extension - Maximum extension of the knee joint at any point in the pedal stroke defined by the line connecting hip and knee markers and the line connecting knee and ankle markers SAW - Shoulder Angle to Wrist - The angle of the shoulder joint defined as the angle at intersection of the line connecting hip and shoulder markers, and the line connecting wrist and shoulder markers BA - Back Angle - The angle of the back relative to the horizon defined by the hip and shoulder marker
pO2_start | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  Mean of first 12s of TcPO₂ measurements in each 10 minute interval.
pO2_end | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  Mean of last 12s of TcPO₂ measurements in each 10 minute interval.
pCO2_start | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  Mean of first 12s of TcPCO₂ measurements in each 10 minute interval.
pCO2_end | During a single laboratory visit consisting of three 10-minute cycling intervals with three 5-minute pause time in between cycling intervals (total assessment time approximately 45 minutes).
  Mean of last 12s of TcPCO₂ measurements in each 10 minute interval.

CONTACTS AND LOCATIONS:
Overall Officials: Milan Martínek, Mgr., Ph.D., Principal Investigator — Charles University, Czech Republic
Locations (1):
- Charles University, Prague, Czechia